CLINICAL TRIAL: NCT04902469
Title: Cognitive and Affective Mechanisms Underlying an Olfactory Approach to Modify Cigarette Craving: A Neurobehavioral Investigation
Brief Title: Cognitive and Affective Mechanisms Underlying an Olfactory Approach to Modify Cigarette Craving
Acronym: OdorCrave
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael A Sayette, PhD, Professor of Psychology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY20070045; R01AT010896-01 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-05-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Craving
Keywords: Craving; Olfaction; mechanistic study
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Intervention Model Description: This is a between-subjects design in which 250 nicotine-deprived smokers, who vary in whether they smoke daily and in motivation to quit, will be exposed to smoking cues to induce peak cravings and then receive either a pleasant (n = 125) or neutral (n = 125) olfactory cue.
Who Masked: Participant
Masking Description: Participants will not be informed about whether they are in the odor blank (control) or pleasant odor (experimental) group. However, the odor blank group is intended to control for the act of sniffing rather than the belief that one has sniffed a pleasant odor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pleasant Odor (Experimental): Participants in this condition will sniff the olfactory cue they rate as both pleasant (>5 on the 1-9 scale) and the most intense following cigarette cue exposure. If this odor is the same as their self-reported preferred e-cigarette flavor, we will choose the next most intense odor out of the odors rated as pleasant.
  Interventions: Behavioral: Pleasant Odor
- Odor Blank (Other): Participants in this condition will sniff a neutral olfactory cue (odor blank) following cigarette cue exposure.
  Interventions: Behavioral: Odor Blank

INTERVENTIONS:
Behavioral: Pleasant Odor — Each participant in the pleasant odor condition will sniff an odor that they rated as the most intense out of a sample of odors rated to be pleasant. If this odor is the same as their self-reported preferred e-cigarette flavor, we will choose the next most intense odor out of the odors rated to be pleasant. Odors are generic and commercially available in supermarkets such as vanilla, coconut, and chocolate. Importantly, the investigators are not testing the specific odors, rather the participant's idiosyncratic response to a menu of odors. In other words, the key is that each participant in the experimental condition receives the odor that they like the best, regardless of which one it is.
  Arms: Pleasant Odor
Behavioral: Odor Blank — Each participant in the odor blank condition will sniff a neutral olfactory cue (odor blank). This involves a container with no added scent. This serves as the control condition.
  Arms: Odor Blank

SUMMARY:
The proposed study uses fMRI and behavioral measures in and outside the laboratory to investigate the neurobehavioral mechanisms underlying the impact of pleasant olfactory cues (OCs) on cigarette craving. The investigators plan to randomize 278 participants to a pleasant OC condition or an odor blank (neutral) condition and due to anticipated drop out expect to run 250 adult (half female) smokers, including both daily and nondaily smokers through the protocol. This study involves three visits. In the first visit, participants will complete a baseline breath carbon monoxide reading, a brief odor threshold test, and complete a series of self-report measures. In the next session, participants who are 8-hrs deprived of nicotine will undergo a 60-minute fMRI scan that will include structural, resting state, and task-based data collection. The fMRI task involves completing a series of tasks designed to index responses linked to key neural networks found to relate to addiction (e.g., reward processing, working memory). Participants will also be exposed to smoking cues to heighten craving and then depending on their condition (randomly assigned) will either receive a pleasant or neutral (odor blank) OC. In the third session, behavioral data will be collected to test the impact of either a pleasant or neutral OC on cigarette craving using self-reported urge and behavioral measures linked to craving. Finally, for pilot purposes designed to offer data for a subsequent clinical study (beyond this study), participants will additionally complete a 7-day ecological momentary assessment (EMA) protocol in which they will monitor cigarette craving and initial data will be collected outside the laboratory to evaluate the impact of OCs on naturally occurring craving. It is hypothesized that pleasant OCs will disrupt craving brain states and attenuate craving (as compared to neutral olfactory cues). Further, it is hypothesized that individual variation in neural responses to cognitive and affective tasks will reveal variation in mechanisms underlying pleasant OC craving reduction and that individual differences will moderate pleasant OC-induced craving relief. Finally, it is also expected that emotional responses to pleasant OCs will mediate the impact of OCs on craving and smoking-related processes.

DETAILED DESCRIPTION:
The investigators aim to conduct a comprehensive analysis of craving and to test the impact of pleasant olfactory cues (OCs) on craving relief. Towards these aims, this study will integrate four sources of data: (a) individual differences thought to relate to craving; (b) neural responses to cognitive tasks and behavioral (e.g., Facial Action Coding System measures) reactions to OC sampling; (c) fMRI and behavioral responses to post-smoking cue OC exposure; and (d) EMA data related to craving and smoking. The investigators will embed findings within neurobehavioral addiction theories (dual-systems, iRISA) and will try to identify individuals who may benefit most from OC-based interventions. Most of the study procedures are observational in that they are intended to measure without influencing any health-related outcome. One study procedure meets the revised NIH guidelines for an intervention, in that craving, behavior, and brain activity are measured while participants are presented with either a pleasant or a neutral (blank) olfactory cue in a between-subjects design. The details of study procedures are outlined in the following paragraphs.

Overview Data will be collected over a series of three laboratory sessions. Nicotine-deprived smokers with varying levels of interest in quitting will sample a set of OCs. Participants will be exposed to smoking cues to induce peak cravings and then receive one of the previous OCs (randomly assigned to either a pleasant or neutral OC). This study will use a between-subjects design in which participants will complete several tasks during two experimental sessions, with some tasks better suited to the behavioral and others to the fMRI session. A week-long EMA protocol will follow, within which the effect of OCs on craving and smoking will be assessed. All participants will complete all study procedures.

Procedures The first study contact includes a telephone screening to assess preliminary inclusion and exclusion criteria, including major MRI-related exclusion criteria such as metal in the body. Eligible and interested participants will then visit the lab to complete an approximately 1-hour visit that includes a standardized assessment. Data collected during this visit will be used primarily to characterize the sample.

In both of the following experimental visits, participants will complete a series of common procedures. First, participants will be asked to abstain from smoking for at least 8-hrs prior to each visit. To ensure abstinence, participants will report when they last used nicotine and record carbon monoxide (CO). Participants will also present their cigarette pack and lighter, and complete a brief assessment of baseline craving and mood with standard measures used in the Principal Investigator's prior work. Additionally, participants undergo an odor sampling procedure. They will be asked to sniff 8 OCs; after each one, they will provide via structured interview ratings of pleasantness, intensity, familiarity, evoked emotions, mood, and report any associations or memories to the OC. OC presentation order is randomized. Participants will then undergo a cigarette cue exposure to induce peak cravings. Participants in the pleasant OC condition will then sniff an OC they rated as pleasant, while those randomized to the neutral condition will receive an odor blank. Outside of these procedures, the two experimental sessions differ.

The first experimental session will occur within approximately 1-week (potentially more depending on scanner availability) of the screening session and will include a roughly 60-minute fMRI scan. The first part of the scan will involve structural, resting state, and task-based data collection (e.g., Go/No-Go to assess response inhibition; cigarette cue exposure). This will allow for identification of individually specified cognitive brain states linked to addiction-related processes (i.e., neural fingerprints). Then, neural activity (BOLD) and functional and effective connectivity for identified regions of interest (ROI) will be measured during a smoking cue exposure manipulation (to induce craving) followed by olfactory cue administration. These data will be used to examine the disruption of the craving brain state by the pleasant, compared to the neutral, olfactory cue.

In the second experimental session, participants will undergo a series of behavioral tasks. This again includes a smoking cue exposure manipulation followed by administration of either the pleasant or neutral olfactory cue. To examine the impact of pleasant vs. neutral OCs on craving, participants will provide urge ratings and behavioral measures of urge (i.e., craving as measured through a pressure-sensitive squeeze device, and facial affect) throughout this procedure. Behavioral measures of affect will also be collected during the OC sampling procedure to allow for an examination of how emotional responses to pleasant olfactory cues mediate the impact of olfactory cues on craving.

The final study procedure involves a 7-day ecological momentary assessment (EMA) protocol in which participants will monitor their cigarette cravings and the investigators will collect pilot data to assess how well pleasant vs. neutral olfactory stimuli will control these real-life cravings.

The primary outcomes of interest throughout these experimental sessions involve the impact of pleasant vs. neutral olfactory cues (i.e., odor blanks) on urge to smoke. The investigators are also interested in determining if the patterns of neural activation during smoking cue exposure and during olfactory cue exposure are more similar for those randomized to the neutral OC condition than to the pleasant OC condition. Briefly, analyses will include representational similarity analysis, in which the similarity of activity patterns (neural fingerprints) for different brain states (craving, post-cigarette cue odor) in each subject, is measured through Pearson correlation. Brain states are represented by the pattern of beta coefficients across the 89 atlas regions that underlie each phase of the fMRI session (e.g., while the subject is holding a cigarette to induce craving). These patterns are correlated with each other (giving one Fisher-Z transformed r coefficient per subject), and the resulting correlation coefficients are compared in a group analysis that tests for a statistically significant difference between the pleasant odor group and the neutral/odor blank group. Secondary outcomes of interest include equivalent analyses that calculate the similarity between the post-cigarette cue odor-induced brain state with brain states observed for each of the behavioral tasks completed in the fMRI ( i.e., N-back, Posner Cueing, Delay Discounting, Go/No-Go) in order to quantify and statistically contrast the relative presence of key cognitive and affective processes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-49
* Right-handed
* Fluent in English
* Intact sense of smell
* Pass an MRI safety screening and along these lines will need to be 250lbs or less to safely enter the MRI
* No drug dependence outside of nicotine or caffeine
* Must fit into one of two categories of smokers, daily or nondaily, as confirmed by verbal self-report and a baseline CO reading; Daily smokers: must smoke 10-30 cigarettes per day for at least 12 months, Nondaily smokers: must smoke for 1-14 days of the last 30 days with no more than 20 cigarettes a day
* Need to have access to a working smartphone to complete the ecological momentary assessment portion of the study

Exclusion Criteria:

* Medical conditions that contraindicate nicotine use
* Not fluent in English
* Illiterate
* Current neurological or psychotic disorders
* Current psychoactive drug use
* MRI contraindications such as stroke history, pregnancy, metal in the body, history of aneurysms, or serious head injury
* Individuals will also be excluded if they report any allergies to the odors used in our study.
* Baseline CO readings will need to be consistent with our criteria for daily and nondaily smokers for participants to be considered eligible. Specifically, we plan to rule out extremely heavy smokers (nondeprived CO > 55, for whom the smoking abstinence requirement may be too extreme to allow a sensitive test of our OC manipulation) and daily smokers with a nondeprived CO reading <10 PPM as this would raise concerns that they do smoke enough to be classified as a daily smoker.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Disruption of the Craving Brain State by the Pleasant, Compared to the Neutral, Olfactory Cue | within 1 month of enrollment; immediately before and after administration of the olfactory cue
  Condition difference in the Fisher Z-transformed correlation coefficient between the craving brain state and olfactory cue-induced brain state, where brain states are indexed as the fMRI contrast between cigarette cue (with, and without, odor) and control cue
Craving Observed During Pleasant Compared to Neutral OC Exposure Assessments, Controlling for Pre-OC Craving Ratings | between 1 and 10 days subsequent to the fMRI study visit; before and immediately after administration of the olfactory cue
  Condition difference in self-reported urge on a 0 to 100 scale, with 0 equal to no urge to smoke at all, and 100 as the "strongest urge to smoke that I have ever felt"

SECONDARY OUTCOMES:
Strength of the Cognitive-Associated Neural Fingerprint Induced During the Pleasant Compared to Neutral Olfactory Cue | within 1 month of enrollment; during the fMRI scan
  The condition difference in Fisher Z-transformed correlation coefficients between each cognitive domain neural fingerprint and olfactory cue-induced brain state
Change in Craving from Peak Craving to the Craving Observed During Pleasant, Compared to Neutral, Olfactory Cues as Measured by a Pressure-Sensitive Squeeze Device | between 1 and 10 days subsequent to the fMRI study visit; immediately before and after administration of the olfactory cue
  Condition difference in behavioral response on a dynamometer pressure-squeeze device, measured as pressure force (intensity x duration)
Mediating Role of the Emotional Response to the Pleasant Olfactory Cue, as Indexed by the Facial Action Coding System, on the Impact of Pleasant Olfactory Cues on Self-Reported Craving | between 1 and 10 days subsequent to the fMRI study visit; immediately before and after administration of the olfactory cue
  Mediating effect of emotional response, as measured by the Duchenne smile in the Facial Action Coding System, on the effect of olfactory cues on self-reported urge, indexed using the 0-100 urge rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Sayette, PhD, Principal Investigator — The University of Pittsburgh; Marc N Coutanche, PhD, Principal Investigator — The University of Pittsburgh
Locations (1):
- The University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Following the publication of research articles featuring data pertaining to this study's specific aims, the investigators will make all participant data (with the exception of facial coding data) and data dictionaries available to users after de-identification. Specifically, de-identified behavioral data and related materials will be made available on the Open Science Foundation. De-identified imaging data will also be uploaded to the Open Science Foundation, and unthresholded fMRI statistical maps will be made publicly available on NeuroVault. Finally, study methods, hypotheses, and primary planned analyses (including the specific region that will be tested in ROI-based analyses) will be pre-registered on the Open Science Framework (OSF) prior to data collection.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study methods, hypotheses, and primary planned analyses will be pre-registered on the Open Science Framework (OSF) prior to data collection. Subsequent to publication of papers based on data pertaining to this investigation's specific aims, de-identified data will be made available for the purposes of research upon access request.
Access Criteria: De-identified study data will be available to researchers who agree to a data-sharing agreement that provides for (1) a commitment to using the data only for noncommercial research purposes and (2) a commitment to securing the data using appropriate computer technology. Unthresholded fMRI statistical maps will be publicly available to all users on NeuroVault.

REFERENCES:
- [Background] Sayette MA, Marchetti MA, Herz RS, Martin LM, Bowdring MA. Pleasant olfactory cues can reduce cigarette craving. J Abnorm Psychol. 2019 May;128(4):327-340. doi: 10.1037/abn0000431. Epub 2019 Apr 15. PMID 30985171
- [Background] Sayette MA, Parrott DJ. Effects of olfactory stimuli on urge reduction in smokers. Exp Clin Psychopharmacol. 1999 May;7(2):151-9. doi: 10.1037//1064-1297.7.2.151. PMID 10340155